CLINICAL TRIAL: NCT02256410
Title: The Effects of a Pain Detecting and Analgesic Stimulating Device on Low Back Pain Patients' Clinical Outcomes
Brief Title: Pain Detecting and Analgesic Stimulating Device on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jo Nijs, Prof. dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeMaLBP
Record Dates: First submitted 2013-12-13; First posted 2014-10-03 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; chronic pain; sensitization; treatment; trigger points
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation (Experimental): Patients will undergo 6 sessions, each including 20 minutes of stimulation. These are given after the Nervomatrix device determines the peak pain regions for each patient, and selects to stimulate the top 10 regions with least skin resistance. The frequency of stimulation is 8Hz, at an intensity matched for each patient's tolerance, without inflicting any pain. The location of the stimulations will change in accordance to the changes in the peak pain regions, reflecting changes in tissue physiology possibly linked to clinical improvements.
  Interventions: Device: Stimulation
- sham stimulation (Sham Comparator): Patients will undergo 6 sessions, each including 20 minutesof sham stimulation (no stimulation). These are given after the Nervomatrix device determines the peak pain regions for each patient, and selects to stimulate the top 10 regions with least skin resistance.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Stimulation — The Nervomatrix device first measures skin impedance, and then creates a digital pain matrix map of the back. Regions with low resistance are then selected for brief electric stimulation, thus targeting the treatment to specific peak pain regions. Preliminary evidence supports the effectiveness of this device in reducing pain and disability over 6 sessions
  Other Names: Nervomatrix
  Arms: Stimulation
Other: Sham — The Nervomatrix device first measures skin impedance, and then creates a digital pain matrix map of the back. Regions with low resistance are then selected for brief mechanical pressure.
  Arms: sham stimulation

SUMMARY:
Purpose of study is to test in a randomized controlled trial (RCT) the effects of the Nervomatrix device on various clinical outcomes of patients with low back pain, as well as its mechanisms of action.

DETAILED DESCRIPTION:
This will be a matched randomized-controlled trial - RCT. Using random numbers from a random number generator, pairs of patients will be randomized to either the Nervomatrix stimulation (experimental group) or to sham stimulation (controls). Matching of pairs will be done based on the baseline data of the primary outcomes - pain and disability, as well as on other treatments received.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain persisting for at least 3 months

Exclusion Criteria:

* patho-anatomical diagnosis (such as fractures, tumors, rheumatic diseases and neurological diseases)
* initiated a new conventional therapy during the study period
* pregnant
* patients having a cardiac pacemaker, implanted defibrillator, or other implanted metallic or electronic device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The change in the amount of steps climbed during one minute | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  Stair climbing: Participants were asked to climb up and down 5 stairs for 1 minute, using the rail for support if required. The total amount of steps climbed will be recorded

SECONDARY OUTCOMES:
The change in central sensitization inventory | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  Part A of 25 statements related to current health symptoms. Each of these items is measured on a 5-point temporal Likert scale, with the following numeric rating scale: never (0), rarely (1), sometimes (2), often (3), and always (4). A cumulative score ranges from 0 to 100. Additionally information is collected in Part B on previously diagnosed central sensitivity syndromes and related conditions.
The change in Pain Catastrophizing Scale | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  will be used to assess pain catastrophizing. It consists of 13 items describing different thoughts and feelings that individuals may experience when they are experiencing pain. Items are scored on a 5-point scale, and total scores are counted by adding up all individual items scores. Higher scores correspond to more severe catastrophic thoughts about pain.
The change in revised Illness perception questionnaire | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  will be used for assessing the patients' illness perceptions, as it is known that patients with maladaptive illness perceptions (e.g. expecting that their back problem will last for a long time, or holding weak beliefs in the controllability of their back problem) are more likely to have poor clinical outcomes 6 months after they consulted their physician
The change in average pain intensity | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  average pain rating in the last seven days using a 100 mm Visual Analogue Scale (VAS)
The change in Quebec Back Pain Disability Scale | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  This questionnaire consists of 20 activity related questions which the patient has to score on a six points scale (0= no; 5= not capable to perform the activity). The total score represents a percentage of functional limitations the patient experiences during daily life.
The change in Tampa Scale of Kinesiophobia | measured prior to the first treatment session (baseline) and immediately following the 6th treatment session (after three weeks)
  Tampa Scale of Kinesiophobia is a 17-item questionnaire developed to measure the fear of movement and (re)injury. Each item is scored on a four-point Likert scale ranging from "strongly disagree" [1] to "strongly agree" [4]. Ratings are added up to give a total score ranging from 17-68 points, with the higher values reflecting greater fear of (re)injury

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium